CLINICAL TRIAL: NCT03221426
Title: A Phase III, Randomized, Double-Blind, Clinical Trial of Pembrolizumab (MK-3475) Plus Chemotherapy (XP or FP) Versus Placebo Plus Chemotherapy (XP or FP) as Neoadjuvant/Adjuvant Treatment for Subjects With Gastric and Gastroesophageal Junction (GEJ) Adenocarcinoma (KEYNOTE-585)
Brief Title: Study of Pembrolizumab (MK-3475) Plus Chemotherapy Versus Placebo Plus Chemotherapy in Participants With Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma (MK-3475-585/KEYNOTE-585)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-585; MK-3475-585 (Other: MSD); 173786 (Registry Identifier: JAPIC); KEYNOTE-585 (Other: MSD); PHRR200226-002534 (Registry Identifier: PHRR Research Registration); 2023-509595-42-00 (Registry Identifier: EU CT); 2016-004408-76 (EudraCT Number)
Record Dates: First submitted 2017-07-17; First posted 2017-07-18 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Stomach Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Saline Solution; Cisplatin; Capecitabine; Fluorouracil; Docetaxel; Oxaliplatin; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pembrolizumab + XP/FP (Experimental): XP=cisplatin+capecitabine and FP=cisplatin+5-fluorouracil. Neoadjuvant: Prior to surgery, participants receive 3 cycles of pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets twice each day (BID) on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 IV infusion on Day 1 Q3W and 5-fluorouracil (5FU) 800 mg/m^2 continuous IV infusion on Days 1 to 5 of each 3-week cycle.
  Adjuvant: 4 to 10 weeks post-surgery, participants receive 3 cycles of pembrolizumab 200 mg IV infusion on Day 1 Q3W PLUS cisplatin 80 mg/m^2 IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets BID on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 IV infusion on Day 1 Q3W and 5FU 800 mg/m^2 continuous IV infusion on Days 1 to 5 of each 3-week cycle, followed by pembrolizumab monotherapy 200 mg IV infusion on Day 1 Q3W for up to 11 additional cycles.
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: Capecitabine; Drug: 5-fluorouracil
- Placebo + XP/FP (Placebo Comparator): Neoadjuvant: Prior to surgery, participants receive 3 cycles of placebo (normal saline solution) via IV infusion on Day 1 Q3W PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets BID on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5FU 800 mg/m^2 via continuous IV infusion on Days 1 to 5 of each 3-week cycle.
  Adjuvant: 4 to 10 weeks post-surgery, participants receive 3 cycles of placebo via IV infusion on Day 1 Q3W PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets BID on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5FU 800 mg/m^2 via continuous IV infusion on Days 1 to 5 of each 3-week cycle, followed by placebo monotherapy via IV infusion on Day 1 Q3W for up to 11 additional cycles.
  Interventions: Drug: Placebo; Drug: Cisplatin; Drug: Capecitabine; Drug: 5-fluorouracil
- Pembrolizumab+FLOT Cohort (Experimental): FLOT=docetaxel+oxaliplatin+5FU+leucovorin (calcium folinate). Neoadjuvant: Prior to surgery, participants receive 3 cycles of pembrolizumab 200 mg via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin (calcium folinate) 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3, for 4 administrations).
  Adjuvant: 4 to 10 weeks postsurgery, participants receive 3 cycles of pembrolizumab 200 mg via IV infusion Day 1 Q3W PLUS docetaxel 50 mg/m^2, oxaliplatin 85 mg/m^2, 5FU 2600 mg/m^2, and leucovorin 200 mg/m^2 Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3, for 4 administrations), followed by pembrolizumab monotherapy 200 mg via IV infusion on Day 1 Q3W for up to 11 additional cycles.
  Interventions: Biological: Pembrolizumab; Drug: 5-fluorouracil; Drug: Docetaxel; Drug: Oxaliplatin; Drug: Leucovorin
- Placebo+FLOT Cohort (Placebo Comparator): Neoadjuvant: Prior to surgery, participants receive 3 cycles of placebo (normal saline solution) via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3, for 4 administrations).
  Adjuvant: 4 to 10 weeks postsurgery, participants receive 3 cycles of placebo via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3, for 4 administrations), followed by placebo monotherapy via IV infusion on Day 1 Q3W for up to 11 additional cycles.
  Interventions: Drug: Placebo; Drug: 5-fluorouracil; Drug: Docetaxel; Drug: Oxaliplatin; Drug: Leucovorin

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + XP/FP; Pembrolizumab+FLOT Cohort
Drug: Placebo — IV infusion
  Other Names: Normal saline solution
  Arms: Placebo + XP/FP; Placebo+FLOT Cohort
Drug: Cisplatin — IV infusion
  Other Names: PLATINOL®
  Arms: Pembrolizumab + XP/FP; Placebo + XP/FP
Drug: Capecitabine — Oral tablets
  Other Names: XELODA®
  Arms: Pembrolizumab + XP/FP; Placebo + XP/FP
Drug: 5-fluorouracil — IV infusion
  Other Names: ADRUCIL®; 5FU
Drug: Docetaxel — IV infusion
  Other Names: TAXOTERE®
  Arms: Pembrolizumab+FLOT Cohort; Placebo+FLOT Cohort
Drug: Oxaliplatin — IV infusion
  Other Names: ELOXATIN®
  Arms: Pembrolizumab+FLOT Cohort; Placebo+FLOT Cohort
Drug: Leucovorin — IV infusion
  Other Names: WELLCOVORIN®
  Arms: Pembrolizumab+FLOT Cohort; Placebo+FLOT Cohort

SUMMARY:
The purpose of this study is to evaluate the efficacy of pembrolizumab (MK-3745) in the neoadjuvant (prior to surgery) or adjuvant (after surgery) treatment of previously untreated adults with gastric and gastroesophageal junction (GEJ) adenocarcinoma.

The primary study hypotheses are that:

* Neoadjuvant and adjuvant pembrolizumab plus chemotherapy, followed by adjuvant pembrolizumab is superior to neoadjuvant and adjuvant placebo plus chemotherapy, followed by adjuvant placebo in terms of Event-free Survival (EFS) based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), and
* Neoadjuvant pembrolizumab plus chemotherapy is superior to neoadjuvant placebo plus chemotherapy in terms of rate of Pathological Complete Response (pathCR) at the time of surgery.

With Amendment 10, upon study completion, participants will be discontinued and may be enrolled in an extension study.

ELIGIBILITY:
Inclusion Criteria:

* Has previously untreated localized gastric or GEJ adenocarcinoma as defined by T3 or greater primary lesion or the presence of any positive nodes - N+ (clinical nodes) without evidence of metastatic disease.
* Plans to proceed to surgery following pre-operative chemotherapy based on standard staging studies per local practice.
* Is willing to provide tissue from a tumor lesion at baseline and at time of surgery.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1 within 3 days prior to the first dose of study treatment.
* Has adequate organ function.
* Male participants of childbearing potential must agree to use an adequate method of contraception for the course of the study through 180 days after the last dose of chemotherapy.
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 180 days after the last dose of chemotherapy or through 120 days after the last dose of pembrolizumab, whichever is greater.
* Has life expectancy of greater than 6 months.

Exclusion Criteria:

* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has received prior therapy with an anti-programmed cell death protein-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (i.e., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], tumor necrosis factor receptor superfamily member 4 [OX-40], necrosis factor receptor superfamily member 9 [CD137]) or has previously participated in a Merck pembrolizumab (MK-3475) clinical trial.
* Has received prior systemic anti-cancer therapy including investigational agents for the current malignancy.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior the first dose of study treatment.
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ that have undergone potentially curative therapy are not excluded.
* Has a known severe hypersensitivity (≥ Grade 3) to pembrolizumab, its active substance and/or any of its excipients, or to any of the study chemotherapy agents and/or to any of their excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of Hepatitis B or known active Hepatitis C virus infection.
* Has a known history of active tuberculosis (TB).
* Female participants who are pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the screening visit through180 days after the last dose of chemotherapy or through 120 days after the last dose of pembrolizumab, whichever is greater.
* Male participants who are expecting to father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of chemotherapy.
* Has had an allogenic tissue/solid organ transplant.
* Has received a live vaccine within 30 days prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1007 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2025-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (171):
- United States (14):
  - City of Hope ( Site 0005), Duarte, California
  - Yale Cancer Center ( Site 0016), New Haven, Connecticut
  - Georgetown University ( Site 0015), Washington D.C., District of Columbia
  - Northwestern University - Robert H. Lurie Comprehensive Cancer Center ( Site 0018), Chicago, Illinois
  - The University of Chicago Medical Center ( Site 0004), Chicago, Illinois
  - Roswell Park Cancer Institute ( Site 0001), Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 0019), New York, New York
  - Memorial Sloan Kettering ( Site 0024), New York, New York
  - Weill Cornell Medical Center ( Site 0023), New York, New York
  - University of Rochester ( Site 0011), Rochester, New York
  - Fox Chase Cancer Center ( Site 0006), Philadelphia, Pennsylvania
  - Temple University Hospital ( Site 0026), Philadelphia, Pennsylvania
  - University of Utah, Huntsman Cancer Institute ( Site 0012), Salt Lake City, Utah
  - Virginia Cancer Specialists, PC ( Site 0010), Fairfax, Virginia
- Belgium (9):
  - Institut Jules Bordet ( Site 0480), Brussels, Bruxelles-Capitale, Region de
  - Hopital Erasme ULB ( Site 0484), Brussels, Bruxelles-Capitale, Region de
  - UCL Saint Luc ( Site 0479), Brussels, Bruxelles-Capitale, Region de
  - Grand Hopital de Charleroi ( Site 0478), Charleroi, Hainaut
  - CHU de Liege ( Site 0482), Liège, Liege
  - CHU UCL Namur Site de Godinne ( Site 0485), Yvoir, Namur
  - UZ Gent ( Site 0486), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0483), Leuven, Vlaams-Brabant
  - AZ Groeninge ( Site 0481), Kortrijk, West-Vlaanderen
- Brazil (8):
  - Instituto do Cancer do Ceara ( Site 0311), Fortaleza, Ceará
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 0308), Porto Alegre, Rio Grande do Sul
  - CEPON - Centro de Pesquisas Oncologicas ( Site 0302), Florianópolis, Santa Catarina
  - Fundacao Pio XII - Hospital de Cancer de Barretos ( Site 0301), Barretos, São Paulo
  - Hospital de Base de Sao Jose de Rio Preto ( Site 0304), Sao Jose Rio Preto, São Paulo
  - Instituto Nacional Do Cancer Jose Alencar Gomes Da Silva ( Site 0307), Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0305), São Paulo
  - Hospital Israelita Albert Einstein ( Site 0309), São Paulo
- Canada (8):
  - Cross Cancer Institute ( Site 0033), Edmonton, Alberta
  - Moncton Hospital - Horizon Health Network ( Site 0038), Moncton, New Brunswick
  - Sunnybrook Research Institute ( Site 0032), Toronto, Ontario
  - CISSS de la Monteregie-Centre ( Site 0039), Greenfield Park, Quebec
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 0040), Montreal, Quebec
  - Jewish General Hospital ( Site 0034), Montreal, Quebec
  - CHU de Quebec - Hotel-Dieu de Quebec ( Site 0042), Québec, Quebec
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0035), Sherbrooke, Quebec
- Chile (5):
  - Hospital Regional Rancagua Libertador Bernardo O Higgins ( Site 0299), Rancagua, Lbtdr Gen Bernardo O Higgins
  - Fundacion Arturo Lopez Perez FALP ( Site 0286), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0285), Santiago, Region M. de Santiago
  - Hospital Clinico Universidad de Chile ( Site 0287), Santiago, Region M. de Santiago
  - Instituto Clinico del Sur. ICOS ( Site 0290), Temuco, Región de la Araucanía
- China (3):
  - Beijing Cancer Hospital ( Site 0221), Beijing, Beijing Municipality
  - Zhejiang Cancer Hospital ( Site 0231), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital ( Site 0233), Hangzhou, Zhejiang
- SA Pohja-Eesti Regionaalhaigla ( Site 0526), Tallinn, Harju, Estonia
- France (12):
  - Hopital Prive Jean Mermoz ( Site 0462), Lyon, Auvergne
  - Institut Paoli Calmettes ( Site 0472), Marseille, Bouches-du-Rhone
  - CHU Reims - Hopital Robert Debre ( Site 0465), Reims, Champagne-Ardenne
  - CHU Brest - Institut de Cancerologie et d Hematologie ( Site 0474), Brest, Finistere
  - CHU Toulouse - Hopital Rangueil ( Site 0470), Toulouse, Haute-Garonne
  - Institut du Cancer de Montpellier ( Site 0473), Montpellier, Herault
  - Centre Eugene Marquis ( Site 0466), Rennes, Ille-et-Vilaine
  - Institut de Cancerologie de l Ouest Centre Rene Gauducheau ( Site 0469), Saint-Herblain, Loire-Atlantique
  - CHRU Lille - Hopital Claude Huriez ( Site 0461), Lille, Nord
  - CHU Poitiers - Pole Regional de Cancerologie ( Site 0467), Poitiers, Vienne
  - CHU Hopital Saint Antoine ( Site 0471), Paris
  - Institut Mutualiste Montsouris ( Site 0463), Paris
- Germany (8):
  - Klinikum Esslingen GmbH ( Site 0453), Esslingen am Neckar, Baden-Wurttemberg
  - Universitaetsklinikum Freiburg ( Site 0450), Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum der Universitaet in Muenchen ( Site 0446), Munich, Bavaria
  - Medizinische Hochschule Hannover ( Site 0449), Hanover, Lower Saxony
  - Kliniken Essen Mitte Gmbh Evang. Huyssens Stiftung ( Site 0445), Essen, North Rhine-Westphalia
  - Medizinische klinilk und Poliklinik Johannes Gutenberg Univ ( Site 0455), Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus der TU Dresden ( Site 0448), Dresden, Saxony
  - Haematologisch-Onkologische Praxis Eppendorf Facharztzentrum Eppendorf - Hope ( Site 0454), Hamburg
- Guatemala (3):
  - Integra Cancer Institute ( Site 0262), Guatemala City
  - Grupo Medico Angeles ( Site 0261), Guatemala City
  - Centro Medico Integral De Cancerología (CEMIC) ( Site 0260), Quetzaltenango
- Israel (7):
  - Meir medical center ( Site 0386), Kfar Saba, Central District
  - Soroka University M.C ( Site 0385), Beersheba, Southern District
  - Sourasky Medical Center. ( Site 0382), Tel Aviv, Tell Abib
  - Rambam Health Care Campus ( Site 0381), Haifa
  - Hadassah Medical Center. Ein Kerem ( Site 0383), Jerusalem
  - Rabin-Medical Center ( Site 0384), Petah Tikva
  - Sheba Medical center ( Site 0387), Ramat Gan
- Italy (7):
  - IRCCS Istituto Oncologico Veneto ( Site 0431), Padova, Abruzzo
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 0430), Milan, Lombardy
  - Istituto Clinico Humanitas Research Hospital ( Site 0432), Rozzano, Milano
  - IRCCS Policlinico San Donato ( Site 0433), San Donato Milanese, Milano
  - Azienda Ospedaliero Universitaria di Modena Policlinico ( Site 0429), Modena
  - Seconda Universita Napoli ( Site 0436), Napoli
  - A.O.U. Santa Maria della Misericordia di Udine ( Site 0434), Udine
- Japan (30):
  - Aichi Cancer Center Hospital ( Site 0165), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0178), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 0186), Matsuyama, Ehime
  - Hokkaido University Hospital ( Site 0160), Sapporo, Hokkaido
  - Hyogo Cancer Center ( Site 0182), Akashi, Hyōgo
  - Kobe University Hospital ( Site 0188), Kobe, Hyōgo
  - Kobe City Medical Center General Hospital ( Site 0181), Kobe, Hyōgo
  - Ibaraki Prefectural Central Hospital ( Site 0177), Kasama, Ibaraki
  - Iwate Medical University Hospital ( Site 0184), Shiwa-gun, Iwate
  - St. Marianna University School of Medicine Hospital ( Site 0187), Kawasaki, Kanagawa
  - Kanagawa Cancer Center ( Site 0167), Yokohama, Kanagawa
  - Kansai Medical University Hospital ( Site 0190), Hirakata, Osaka
  - Osaka University Hospital ( Site 0162), Suita, Osaka
  - Osaka Medical College Hospital ( Site 0168), Takatsuki, Osaka
  - Saitama Cancer Center ( Site 0170), Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center Hospital and Research Institute ( Site 0176), Sunto-gun, Shizuoka
  - Chiba Cancer Center ( Site 0180), Chiba
  - National Hospital Organization Kyushu Cancer Center ( Site 0172), Fukuoka
  - Kyushu University Hospital ( Site 0173), Fukuoka
  - Gifu University Hospital ( Site 0166), Gifu
  - Hiroshima City Hiroshima Citizens Hospital ( Site 0171), Hiroshima
  - Kochi Health Sciences Center ( Site 0189), Kochi
  - Kumamoto University Hospital ( Site 0164), Kumamoto
  - Niigata Cancer Center Hospital ( Site 0169), Niigata
  - Osaka International Cancer Institute ( Site 0161), Osaka
  - Osaka General Medical Center ( Site 0159), Osaka
  - National Cancer Center Hospital ( Site 0179), Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 0183), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 0185), Tokyo
  - Toyama Prefectural Central Hospital ( Site 0163), Toyama
- Riga East Clinical University Hospital ( Site 0550), Riga, Latvia
- Lithuania (3):
  - LSMUL Kauno Klinikos ( Site 0570), Kaunas
  - Nacionalinis Vezio Institutas ( Site 0569), Vilnius
  - Vilniaus Universiteto Ligonine Santaros Klinikos ( Site 0568), Vilnius
- Malaysia (2):
  - Hospital Kuala Lumpur ( Site 0146), Kuala Lumpur
  - University Malaya Medical Centre ( Site 0143), Kuala Lumpur
- St. Luke s Medical Center ( Site 0622), Quezon City, National Capital Region, Philippines
- Poland (9):
  - Szpital Uniwersytecki w Krakowie ( Site 0352), Krakow, Lesser Poland Voivodeship
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu ( Site 0358), Wroclaw, Lower Silesian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie ( Site 0351), Lublin, Lublin Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 0349), Warsaw, Masovian Voivodeship
  - Mazowiecki Szpital Onkologiczny ( Site 0363), Wieliszew, Masovian Voivodeship
  - Szpital Specjalistyczny w Koscierzynie Sp. z o.o. ( Site 0353), Kościerzyna, Pomeranian Voivodeship
  - Beskidzkie Centrum Onkologii im. Jana Pawla II ( Site 0354), Bielsko-Biala, Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 0361), Gliwice, Silesian Voivodeship
  - SPZOZ WSS nr 3 w Rybniku ( Site 0357), Rybnik, Silesian Voivodeship
- Russia (8):
  - Kaluga Regional Clinical Oncology Center ( Site 0345), Kaluga, Kaluzskaja Oblast
  - SBHI Leningrad Regional Clinical Hospital ( Site 0496), Saint Petersburg, Leningradskaya Oblast'
  - National Medical and Surgical Center n.a. N.I.Pirogov ( Site 0338), Moscow, Moscow
  - Blokhin National Medical Oncology ( Site 0494), Moscow, Moscow
  - Leningrad Regional Oncology Center ( Site 0335), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 0344), Saint Petersburg, Sankt-Peterburg
  - City clinical oncological dispensary ( Site 0336), Saint Petersburg, Sankt-Peterburg
  - Tomsk Scientific Research Institute of Oncology ( Site 0337), Tomsk, Tomsk Oblast
- Singapore (3):
  - National University Hospital ( Site 0095), Singapore, Central Singapore
  - National Cancer Centre Singapore ( Site 0097), Singapore, Central Singapore
  - Oncocare Cancer Centre ( Site 0096), Singapore, Central Singapore
- South Korea (10):
  - Chonnam National University Hwasun Hospital ( Site 0083), Hwasun Gun, Jeonranamdo
  - Seoul National University Bundang Hospital ( Site 0085), Seongnam-si, Kyonggi-do
  - Kyungpook National University Chilgok Hospital ( Site 0089), Daegu, Taegu-Kwangyokshi
  - Gachon University Gil Medical Center ( Site 0087), Incheon
  - Korea University Anam Hospital ( Site 0084), Seoul
  - Seoul National University Hospital -SNUH- ( Site 0080), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0081), Seoul
  - Asan Medical Center ( Site 0082), Seoul
  - Gangnam Severance Hospital ( Site 0088), Seoul
  - SMG-SNU BORAMAE Medical Center ( Site 0086), Seoul
- Taiwan (6):
  - Taipei Medical University Shuang Ho Hospital ( Site 0068), New Taipei City
  - National Cheng Kung University Hospital ( Site 0067), Tainan
  - National Taiwan University Hospital ( Site 0063), Taipei
  - Mackay Memorial Hospital ( Site 0065), Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 0066), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 0064), Taoyuan District
- Ukraine (6):
  - City Clinical Hosp.4 of DCC ( Site 0325), Dnipro, Dnipropetrovsk Oblast
  - MI Kryvyi Rih Oncology Dispensary of Dnipropetrovsk Regional Council ( Site 0589), Kryviy Rih, Dnipropetrovsk Oblast
  - Ivano-Frankivsk Regional Oncology Clinical Dispensary ( Site 0321), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Communal non profit enterprise Regional Clinical Oncology Center ( Site 0591), Kharkiv, Kharkivs’ka Oblast’
  - National Cancer Institute of the MoH of Ukraine ( Site 0319), Kyiv, Kyivska Oblast
  - Kyiv City Clinical Oncology Center ( Site 0590), Kyiv, Kyivska Oblast
- United Kingdom (7):
  - University Hospitals Bristol NHS Foundation Trust ( Site 0407), Bristol, Bristol, City of
  - Ninewells Hospital and Medical School ( Site 0406), Dundee, Dundee City
  - Royal Free London NHS Foundation Trust ( Site 0403), London, London, City of
  - The Royal Marsden Foundation Trust ( Site 0405), London, London, City of
  - Imperial College Healthcare NHS Trust ( Site 0402), London, London, City of
  - Royal Marsden NHS Foundation Trust ( Site 0400), Sutton, Surrey
  - The Christie NHS Foundation Trust ( Site 0397), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Shitara K, Rha SY, Wyrwicz LS, Oshima T, Karaseva N, Osipov M, Yasui H, Yabusaki H, Afanasyev S, Park YK, Al-Batran SE, Yoshikawa T, Yanez P, Dib Bartolomeo M, Lonardi S, Tabernero J, Van Cutsem E, Janjigian YY, Oh DY, Xu J, Fang X, Shih CS, Bhagia P, Bang YJ; KEYNOTE-585 investigators. Neoadjuvant and adjuvant pembrolizumab plus chemotherapy in locally advanced gastric or gastro-oesophageal cancer (KEYNOTE-585): an interim analysis of the multicentre, double-blind, randomised phase 3 study. Lancet Oncol. 2024 Feb;25(2):212-224. doi: 10.1016/S1470-2045(23)00541-7. Epub 2023 Dec 19. PMID 38134948
- [Derived] Shitara K, Rha SY, Wyrwicz L, Oshima T, Karaseva N, Osipov M, Yasui H, Yabusaki H, Afanasyev S, Park YK, Al-Batran SE, Yoshikawa T, Yanez P, Pietrantonio F, Lonardi S, Fang X, Guan Y, Valderrama A, Leconte P, Bhagia P, Bang YJ; KEYNOTE-585 Investigators. Pembrolizumab Plus Chemotherapy Versus Chemotherapy as Perioperative Therapy in Locally Advanced Gastric and Gastroesophageal Junction Cancer: Final Analysis of the Randomized, Phase III KEYNOTE-585 Study. J Clin Oncol. 2025 Oct 10;43(29):3152-3159. doi: 10.1200/JCO-25-00486. Epub 2025 Aug 19. PMID 40829093
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069
- [Derived] Bang YJ, Van Cutsem E, Fuchs CS, Ohtsu A, Tabernero J, Ilson DH, Hyung WJ, Strong VE, Goetze TO, Yoshikawa T, Tang LH, Hwang PMT, Webb N, Adelberg D, Shitara K. KEYNOTE-585: Phase III study of perioperative chemotherapy with or without pembrolizumab for gastric cancer. Future Oncol. 2019 Mar;15(9):943-952. doi: 10.2217/fon-2018-0581. Epub 2019 Feb 19. PMID 30777447
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26112&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1007 participants that were randomized to trial, 1001 received treatment. At the time of the primary analysis data cut-off, 521 participants are ongoing in the study. Analysis of the remaining 521 enrolled participants will be included in the End of Trial analysis.
Groups:
- Pembrolizumab + XP/FP: XP=cisplatin+capecitabine and FP=cisplatin+5-fluorouracil. Neoadjuvant: Prior to surgery, participants receive 3 cycles of pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets twice each day (BID) on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5-fluorouracil (5FU) 800 mg/m^2 via continuous IV infusion on Days 1 to 5 of each 3-week cycle.
  Adjuvant: 4 to 10 weeks post-surgery, participants receive 3 cycles of pembrolizumab 200 mg via IV infusion on Day 1 Q3W PLUS cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and capecitabine 1000 mg/m^2 via oral tablets BID on Days 1 to 14 of each 3-week cycle OR cisplatin 80 mg/m^2 via IV infusion on Day 1 Q3W and 5FU 800 mg/m^2 via continuous IV infusion on Days 1 to 5 of each 3-week cycle, followed by pembrolizumab monotherapy 200 mg via IV infusion on Day 1 Q3W for up to 11 additional cycles.
- Pembrolizumab + FLOT Cohort: FLOT=docetaxel+oxaliplatin+5FU+leucovorin (calcium folinate). Neoadjuvant: Prior to surgery, participants receive 3 cycles of pembrolizumab 200 mg via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin (calcium folinate) 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3, for 4 administrations).
  Adjuvant: 4 to 10 weeks post-surgery, participants receive 3 cycles of pembrolizumab 200 mg via IV infusion Day 1 Q3W PLUS docetaxel 50 mg/m^2, oxaliplatin 85 mg/m^2, 5FU 2600 mg/m^2, and leucovorin 200 mg/m^2 Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3, for 4 administrations), followed by pembrolizumab monotherapy 200 mg via IV infusion on Day 1 Q3W for up to 11 additional cycles.
- Placebo + FLOT Cohort: Neoadjuvant: Prior to surgery, participants receive 3 cycles of placebo (normal saline solution) via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3, for 4 administrations).
  Adjuvant: 4 to 10 weeks post-surgery, participants receive 3 cycles of placebo via IV infusion on Day 1 Q3W PLUS docetaxel 50 mg/m^2 via IV infusion, oxaliplatin 85 mg/m^2 via IV infusion, 5FU 2600 mg/m^2 via IV infusion, and leucovorin 200 mg/m^2 via IV infusion Q2W (on Days 1 and 15 of Cycle 1; Day 8 of Cycle 2, and Day 1 of Cycle 3, for 4 administrations), followed by placebo monotherapy via IV infusion on Day 1 Q3W for up to 11 additional cycles.
Period: Overall Study
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP | Pembrolizumab + FLOT Cohort | Placebo + FLOT Cohort
Started | 402 | 402 | 100 | 103
Treated | 399 | 400 | 99 | 103
Completed | 0 | 0 | 0 | 0
Not Completed | 402 | 402 | 100 | 103
Not completed — Ongoing in study | 212 | 193 | 61 | 55
Not completed — Withdrawal by Subject | 12 | 4 | 2 | 3
Not completed — Lost to Follow-up | 4 | 1 | 1 | 0
Not completed — Death | 174 | 204 | 36 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP | Pembrolizumab + FLOT Cohort | Placebo + FLOT Cohort | Total
Number analyzed (Participants) | 402 | 402 | 100 | 103 | 1007
Age, Customized [Count of Participants; unit: Participants]
  Adults (between 18 and 64 years) | 207 | 221 | 58 | 64 | 550
  From 65 to 84 years | 194 | 181 | 42 | 39 | 456
  85 years and older | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 115 | 22 | 32 | 283
  Male | 288 | 287 | 78 | 71 | 724
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 56 | 11 | 9 | 120
  Not Hispanic or Latino | 333 | 321 | 89 | 94 | 837
  Unknown or Not Reported | 25 | 25 | 0 | 0 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 194 | 193 | 4 | 4 | 395
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 1 | 2 | 11
  White | 178 | 174 | 92 | 97 | 541
  More than one race | 5 | 7 | 2 | 0 | 14
  Unknown or Not Reported | 22 | 23 | 0 | 0 | 45
Geographic Region [Count of Participants; unit: Participants] — Participants were categorized according to geographic region of site: Asia, Western Europe, United States (US), and Rest of World (ROW).
  Participants
    Asia | 190 | 191 | 3 | 3 | 387
    US | 3 | 6 | 9 | 7 | 25
    Western Europe | 104 | 95 | 56 | 70 | 325
    ROW | 105 | 110 | 32 | 23 | 270
Tumor Staging [Count of Participants; unit: Participants] — Participants were categorized by tumor stage based on American Joint Committee on Cancer (AJCC) staging guidelines. The lower the cancer stage, the less the cancer has spread. Stages can range from I to IVd. 'a' describes less aggressive (slower growing) cancer, while 'd' describes more aggressive (faster growing) cancer within a numeric stage.
  Participants
    Stage II | 82 | 80 | 22 | 31 | 215
    Stage III | 302 | 306 | 74 | 66 | 748
    Stage IVa | 18 | 15 | 4 | 6 | 43
    Missing | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) Per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms
Description: EFS is based on RECIST 1.1 as assessed by the investigator and is defined as the time from randomization to the first of the following events: radiographic disease progression per RECIST 1.1; local or distant recurrence as assessed by computer tomography (CT) scan or biopsy if indicated (for participants who are disease free after surgery); clinical progression as evidenced by peritoneal carcinomatosis confirmed by preoperative laparoscopy or laparotomy (for participants who are confirmed to be free of peritoneal involvement by laparoscopy at screening); or death due to any cause. A second primary malignancy, or radiographic progressive disease (PD) during the neoadjuvant phase that does not preclude successful surgery (i.e., disease free after surgery), are not considered EFS events.
Time Frame: Up to approximately 75 months
Population: The analysis population consisted of all randomized participants in the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms, as pre-specified per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP
Number analyzed (Participants) | 402 | 402
Months | 44.4 [33.0 to 69.8] | 25.7 [20.8 to 36.5]
Statistical Analysis 1: Comparison: Pembrolizumab + XP/FP vs Placebo + XP/FP; Test type: Superiority; p = 0.01501, Log Rank — One-sided p-value based on log-rank test stratified by geographic region (Asia vs. Non-Asia) and tumor staging (II vs. III vs. IVa); Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.67 to 0.98] — Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region (Asia vs. Non-Asia) and tumor staging (II vs. III vs. IVa)

2. Primary Outcome: Pathological Complete Response (pathCR) Rate - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms
Description: PathCR rate is defined as the percentage of participants having a pathCR based on central review. pathCR is defined as no invasive disease within an entirely submitted and evaluated gross lesion, and histologically negative nodes. The percentage of participants having pathCR is presented for the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms.
Time Frame: Up to approximately 9 weeks following completion of neoadjuvant treatment (up to Study Week 18)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP
Number analyzed (Participants) | 402 | 402
Percentage of Participants | 13.4 [10.3 to 17.2] | 2.0 [0.9 to 3.9]
Statistical Analysis 1: Comparison: Pembrolizumab + XP/FP vs Placebo + XP/FP; Test type: Superiority; p < 0.00001, Stratified Miettinen and Nurminen; Based on Miettinen & Nurminen method stratified by geographic region (Asia vs. Non-Asia) and tumor staging (II vs. III vs. IVa); Difference in Percentage = 11.4, 95% CI 2-sided [8.0 to 15.3]

3. Primary Outcome: Overall Survival (OS) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms
Description: OS is defined as the time from randomization to death due to any cause. OS is presented for the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms.
Time Frame: Up to approximately 75 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP
Number analyzed (Participants) | 402 | 402
Months | 71.8 [52.5 to NA] — NA = Upper limit was not reached at time of data cut-off due to insufficient number of participants with an event | 55.7 [41.7 to NA] — NA = Upper limit was not reached at time of data cut-off due to insufficient number of participants with an event
Statistical Analysis 1: Comparison: Pembrolizumab + XP/FP vs Placebo + XP/FP; Test type: Superiority; p = 0.07503, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.71 to 1.06] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs) - Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE is presented for the Pembrolizumab+FLOT and Placebo+FLOT Cohorts.
Time Frame: Up to approximately 70 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment in the Pembrolizumab+FLOT and Placebo+FLOT Cohort treatment arms, as pre-specified per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + FLOT Cohort | Placebo + FLOT Cohort
Number analyzed (Participants) | 99 | 103
Participants | 99 | 103

5. Primary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE - Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinued study treatment due to an AE is presented for the Pembrolizumab+FLOT and Placebo+FLOT Cohorts.
Time Frame: Up to approximately 17 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + FLOT Cohort | Placebo + FLOT Cohort
Number analyzed (Participants) | 99 | 103
Participants | 37 | 26

6. Secondary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms Separately and in Combination With the Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience at least one AE will be presented for the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms separately and in combination with the Pembrolizumab+FLOT and Placebo+FLOT Cohorts.
Time Frame: Up to approximately 75 months
Reporting Status: Not Posted, anticipated posting 2026-05

7. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms Separately and in Combination With the Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be presented the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms separately and in combination with the Pembrolizumab+FLOT and Placebo+FLOT Cohorts.
Time Frame: Up to approximately 18 months
Reporting Status: Not Posted, anticipated posting 2026-05

8. Secondary Outcome: Disease-free Survival (DFS) Per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms
Description: DFS is defined as the time from post-surgery baseline scan until the first occurrence of local or distant recurrence or death from any cause and is based on RECIST 1.1 as assessed by the investigator.
Time Frame: Up to approximately 75 months
Population: The analysis population consisted of all randomized participants in the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms who had surgery, as pre-specified per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP
Number analyzed (Participants) | 320 | 306
Months | 66.1 [44.9 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event | 44.2 [27.6 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event
Statistical Analysis 1: Comparison: Pembrolizumab + XP/FP vs Placebo + XP/FP; Test type: Other; p = 0.04125, Log Rank — One-sided p-value based on log-rank test with stratification; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.65 to 1.03] — Cox regression model with Efron's method of tie handling with treatment as a covariate with stratification

9. Secondary Outcome: Overall Survival (OS) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms in Combination With the Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: OS is defined as the time from randomization to death due to any cause. OS is presented for the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms in combination with the Pembrolizumab+FLOT and Placebo+FLOT Cohorts.
Time Frame: Up to approximately 75 months
Population: The analysis population consisted of all randomized participants in the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms in combination with the Pembrolizumab+FLOT and Placebo+FLOT Cohorts, as pre-specified in the protocol.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined: Neoadjuvant and adjuvant pembrolizumab+XP/FP and neoadjuvant and adjuvant pembrolizumab+FLOT Cohort treatment arms combined
- Placebo + XP/FP and Placebo + FLOT Cohort Combined: Neoadjuvant and adjuvant placebo+XP/FP and neoadjuvant and adjuvant placebo+FLOT Cohort treatment arms combined
Arm/Group | Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined | Placebo + XP/FP and Placebo + FLOT Cohort Combined
Number analyzed (Participants) | 502 | 505
Months | NA [59.2 to NA] — NA = Median and upper limit were not reached at the data cut-off due to insufficient number of participants with an event | 55.7 [42.8 to NA] — NA = Upper limit was not reached at the data cut-off due to insufficient number of participants with an event
Statistical Analysis 1: Comparison: Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined vs Placebo + XP/FP and Placebo + FLOT Cohort Combined; Test type: Superiority; p = 0.04493, Log Rank — One-sided p-value based on log-rank test stratified by geographic region (Asia vs. Non-Asia), tumor staging (II vs. III vs. IVa), and chemotherapy backbone (XP/FP vs. FLOT); Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.71 to 1.03] — Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by geographic region (Asia vs. Non-Asia), tumor staging (II vs. III vs. IVa), and chemotherapy backbone (XP/FP vs. FLOT)

10. Secondary Outcome: Event-free Survival (EFS) Per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) - Pembrolizumab+XP/FP and Placebo+XP/FP Treatment Arms in Combination With the Pembrolizumab+FLOT and Placebo+FLOT Cohorts
Description: EFS is based on RECIST 1.1 as assessed by the investigator and is defined as the time from randomization to the first of the following events: radiographic disease progression per RECIST 1.1; local or distant recurrence as assessed by CT scan or biopsy if indicated (for participants who are disease free after surgery); clinical progression as evidenced by peritoneal carcinomatosis confirmed by preoperative laparoscopy or laparotomy (for participants who are confirmed to be free of peritoneal involvement by laparoscopy at screening); or death due to any cause. A second primary malignancy, or radiographic progressive disease (PD) during the neoadjuvant phase that does not preclude successful surgery (i.e., disease free after surgery), are not considered EFS events.
Time Frame: Up to approximately 75 months
Population: The analysis population consisted of all randomized participants in the Pembrolizumab+XP/FP and Placebo+XP/FP treatment arms in combination with the Pembrolizumab+FLOT and Placebo+FLOT Cohorts, as pre-specified per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined: Neoadjuvant and adjuvant pembrolizumab + XP/FP and neoadjuvant and adjuvant pembrolizumab + FLOT Cohort treatment arms combined
Arm/Group | Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined | Placebo + XP/FP and Placebo + FLOT Cohort Combined
Number analyzed (Participants) | 502 | 505
Months | 47.0 [36.2 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event | 26.9 [22.1 to 34.7]
Statistical Analysis 1: Comparison: Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined vs Placebo + XP/FP and Placebo + FLOT Cohort Combined; Test type: Superiority; p = 0.00589, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.67 to 0.95] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to approximately 75 months
Description: All-Cause Mortality includes all randomized participants. Serious and Other adverse events (AEs) includes all randomized participants who received ≥1 dose of study treatment. MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. Per protocol, AEs are presented for the XP/FP and FLOT treatment arms separately and in combination.
Arm/Group | Pembrolizumab + XP/FP | Placebo + XP/FP | Pembrolizumab + FLOT Cohort | Placebo + FLOT Cohort | Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined | Placebo + XP/FP and Placebo + FLOT Cohort Combined
All-Cause Mortality (participants affected / at risk) | 181/402 | 206/402 | 37/100 | 47/103 | 218/502 | 253/505
Serious Adverse Events (participants affected / at risk) | 176/399 | 161/400 | 66/99 | 51/103 | 242/498 | 212/503
Other Adverse Events (participants affected / at risk) | 392/399 | 392/400 | 99/99 | 103/103 | 491/498 | 495/503
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + XP/FP (N=399) | Placebo + XP/FP (N=400) | Pembrolizumab + FLOT Cohort (N=99) | Placebo + FLOT Cohort (N=103) | Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined (N=498) | Placebo + XP/FP and Placebo + FLOT Cohort Combined (N=503)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 6 (6) | 0 (0) | 0 (0) | 5 (5) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 12 (12) | 5 (5) | 6 (6) | 8 (8) | 18 (18)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Toxic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 7 (8) | 2 (2) | 2 (2) | 4 (4) | 9 (10)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 11 (12) | 3 (3) | 1 (1) | 4 (5) | 12 (13) | 7 (8)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 10 (12) | 6 (6) | 2 (2) | 12 (12) | 12 (14)
Dumping syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 4 (5) | 3 (3) | 0 (0) | 5 (5) | 4 (5)
Enteritis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Fistula of small intestine (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Gastric stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 3 (3)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 2 (2) | 2 (2) | 1 (2) | 3 (4) | 3 (4)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 7 (8) | 1 (1) | 2 (2) | 6 (7) | 9 (10)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Omental infarction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Terminal ileitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 9 (11) | 9 (10) | 7 (7) | 2 (2) | 16 (18) | 11 (12)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (5) | 3 (3) | 0 (0) | 1 (1) | 3 (5) | 4 (4)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Physical deconditioning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 5 (6) | 7 (10) | 2 (2) | 11 (14) | 7 (8)
Serositis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hepatic ischaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 6 (6) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abscess soft tissue (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 4 (4)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 6 (6) | 2 (2)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Mediastinal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8) | 4 (5) | 5 (6) | 3 (3) | 13 (14) | 7 (8)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyopneumothorax (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 4 (4) | 3 (3) | 1 (1) | 7 (7) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stoma site abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Afferent loop syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anastomotic fistula (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 4 (4) | 4 (4)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drain site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to anastomose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 3 (3) | 4 (4) | 7 (7) | 5 (5)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Glaucoma traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pancreatic leak (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Escherichia test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (5) | 4 (4) | 0 (0) | 0 (0) | 4 (5) | 4 (4)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (10) | 14 (15) | 2 (2) | 0 (0) | 11 (12) | 14 (15)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 5 (5) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6) | 1 (1) | 1 (1) | 5 (5) | 7 (7)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alcoholic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 3 (3)
Thrombotic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 4 (4)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal salt-wasting syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mediastinal effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 7 (7) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5) | 2 (2) | 2 (2) | 10 (10) | 7 (7)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Embolism (Vascular disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 6 (6) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Internal haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + XP/FP (N=399) | Placebo + XP/FP (N=400) | Pembrolizumab + FLOT Cohort (N=99) | Placebo + FLOT Cohort (N=103) | Pembrolizumab + XP/FP and Pembrolizumab + FLOT Cohort Combined (N=498) | Placebo + XP/FP and Placebo + FLOT Cohort Combined (N=503)
Anaemia (Blood and lymphatic system disorders) | 170 (237) | 159 (213) | 26 (49) | 26 (49) | 196 (286) | 185 (262)
Leukopenia (Blood and lymphatic system disorders) | 16 (27) | 23 (37) | 5 (5) | 5 (6) | 21 (32) | 28 (43)
Neutropenia (Blood and lymphatic system disorders) | 114 (198) | 111 (192) | 27 (44) | 23 (36) | 141 (242) | 134 (228)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (22) | 26 (32) | 4 (6) | 7 (9) | 23 (28) | 33 (41)
Tachycardia (Cardiac disorders) | 3 (3) | 2 (2) | 5 (5) | 3 (4) | 8 (8) | 5 (6)
Tinnitus (Ear and labyrinth disorders) | 29 (30) | 29 (36) | 1 (1) | 0 (0) | 30 (31) | 29 (36)
Hyperthyroidism (Endocrine disorders) | 14 (15) | 5 (5) | 6 (7) | 5 (5) | 20 (22) | 10 (10)
Hypothyroidism (Endocrine disorders) | 35 (37) | 10 (10) | 7 (8) | 5 (5) | 42 (45) | 15 (15)
Abdominal pain (Gastrointestinal disorders) | 58 (101) | 67 (90) | 24 (37) | 31 (54) | 82 (138) | 98 (144)
Abdominal pain upper (Gastrointestinal disorders) | 20 (20) | 30 (31) | 10 (13) | 15 (17) | 30 (33) | 45 (48)
Constipation (Gastrointestinal disorders) | 109 (153) | 111 (150) | 22 (30) | 32 (44) | 131 (183) | 143 (194)
Diarrhoea (Gastrointestinal disorders) | 149 (221) | 131 (206) | 69 (145) | 75 (175) | 218 (366) | 206 (381)
Dry mouth (Gastrointestinal disorders) | 11 (13) | 10 (13) | 7 (8) | 4 (5) | 18 (21) | 14 (18)
Dyspepsia (Gastrointestinal disorders) | 39 (60) | 30 (39) | 5 (5) | 11 (12) | 44 (65) | 41 (51)
Dysphagia (Gastrointestinal disorders) | 21 (23) | 21 (22) | 10 (12) | 12 (12) | 31 (35) | 33 (34)
Flatulence (Gastrointestinal disorders) | 7 (7) | 5 (5) | 6 (7) | 6 (6) | 13 (14) | 11 (11)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 18 (20) | 16 (16) | 9 (9) | 13 (14) | 27 (29) | 29 (30)
Nausea (Gastrointestinal disorders) | 240 (465) | 246 (500) | 58 (109) | 61 (111) | 298 (574) | 307 (611)
Stomatitis (Gastrointestinal disorders) | 63 (82) | 52 (68) | 14 (16) | 9 (11) | 77 (98) | 61 (79)
Vomiting (Gastrointestinal disorders) | 102 (169) | 109 (177) | 38 (62) | 44 (73) | 140 (231) | 153 (250)
Asthenia (General disorders) | 87 (155) | 75 (119) | 20 (29) | 20 (27) | 107 (184) | 95 (146)
Chest pain (General disorders) | 7 (9) | 9 (11) | 5 (5) | 5 (9) | 12 (14) | 14 (20)
Chills (General disorders) | 3 (3) | 5 (6) | 12 (16) | 7 (8) | 15 (19) | 12 (14)
Fatigue (General disorders) | 89 (135) | 92 (127) | 57 (76) | 55 (89) | 146 (211) | 147 (216)
Malaise (General disorders) | 36 (52) | 42 (65) | 0 (0) | 2 (2) | 36 (52) | 44 (67)
Mucosal inflammation (General disorders) | 25 (32) | 25 (32) | 10 (12) | 9 (9) | 35 (44) | 34 (41)
Oedema peripheral (General disorders) | 19 (21) | 19 (24) | 9 (12) | 10 (14) | 28 (33) | 29 (38)
Pyrexia (General disorders) | 65 (79) | 56 (68) | 25 (43) | 26 (34) | 90 (122) | 82 (102)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 5 (5) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 5 (5) | 4 (4) | 8 (8) | 6 (6)
Oral candidiasis (Infections and infestations) | 4 (4) | 4 (5) | 5 (5) | 4 (8) | 9 (9) | 8 (13)
Pneumonia (Infections and infestations) | 13 (14) | 13 (13) | 5 (6) | 5 (5) | 18 (20) | 18 (18)
Urinary tract infection (Infections and infestations) | 7 (7) | 13 (16) | 6 (6) | 9 (9) | 13 (13) | 22 (25)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 6 (6) | 7 (7) | 8 (9) | 8 (8)
Procedural pain (Injury, poisoning and procedural complications) | 37 (37) | 36 (37) | 4 (4) | 4 (4) | 41 (41) | 40 (41)
Wound complication (Injury, poisoning and procedural complications) | 25 (28) | 26 (27) | 0 (0) | 1 (1) | 25 (28) | 27 (28)
Alanine aminotransferase increased (Investigations) | 27 (42) | 26 (36) | 17 (22) | 13 (20) | 44 (64) | 39 (56)
Aspartate aminotransferase increased (Investigations) | 30 (43) | 24 (35) | 15 (20) | 13 (21) | 45 (63) | 37 (56)
Blood alkaline phosphatase increased (Investigations) | 9 (11) | 10 (11) | 8 (9) | 6 (8) | 17 (20) | 16 (19)
Blood creatinine increased (Investigations) | 56 (77) | 53 (88) | 5 (5) | 1 (1) | 61 (82) | 54 (89)
Neutrophil count decreased (Investigations) | 146 (297) | 130 (244) | 40 (83) | 34 (90) | 186 (380) | 164 (334)
Platelet count decreased (Investigations) | 46 (82) | 60 (89) | 11 (24) | 12 (30) | 57 (106) | 72 (119)
Weight decreased (Investigations) | 108 (111) | 104 (111) | 38 (41) | 28 (30) | 146 (152) | 132 (141)
White blood cell count decreased (Investigations) | 69 (145) | 53 (110) | 18 (32) | 15 (31) | 87 (177) | 68 (141)
Decreased appetite (Metabolism and nutrition disorders) | 160 (259) | 169 (252) | 39 (56) | 34 (43) | 199 (315) | 203 (295)
Dehydration (Metabolism and nutrition disorders) | 13 (13) | 11 (12) | 8 (10) | 6 (7) | 21 (23) | 17 (19)
Hyperglycaemia (Metabolism and nutrition disorders) | 15 (17) | 12 (14) | 5 (5) | 7 (9) | 20 (22) | 19 (23)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 (26) | 18 (23) | 8 (9) | 7 (9) | 29 (35) | 25 (32)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (10) | 6 (7) | 6 (6) | 4 (5) | 13 (16) | 10 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 38 (52) | 48 (59) | 11 (18) | 18 (31) | 49 (70) | 66 (90)
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 (15) | 17 (20) | 12 (14) | 3 (3) | 26 (29) | 20 (23)
Hyponatraemia (Metabolism and nutrition disorders) | 13 (22) | 20 (23) | 5 (5) | 5 (9) | 18 (27) | 25 (32)
Hypophosphataemia (Metabolism and nutrition disorders) | 12 (13) | 8 (9) | 8 (8) | 3 (3) | 20 (21) | 11 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (25) | 18 (19) | 15 (20) | 13 (13) | 38 (45) | 31 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (21) | 21 (23) | 9 (12) | 13 (14) | 27 (33) | 34 (37)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 8 (9) | 4 (8) | 9 (10) | 5 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5) | 9 (9) | 2 (2) | 16 (16) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (13) | 15 (16) | 6 (6) | 4 (6) | 16 (19) | 19 (22)
Dizziness (Nervous system disorders) | 34 (39) | 36 (46) | 9 (12) | 12 (14) | 43 (51) | 48 (60)
Dysgeusia (Nervous system disorders) | 45 (52) | 39 (47) | 13 (16) | 12 (15) | 58 (68) | 51 (62)
Headache (Nervous system disorders) | 29 (39) | 30 (39) | 17 (22) | 11 (12) | 46 (61) | 41 (51)
Neuropathy peripheral (Nervous system disorders) | 20 (24) | 25 (25) | 20 (21) | 28 (31) | 40 (45) | 53 (56)
Paraesthesia (Nervous system disorders) | 9 (10) | 11 (15) | 19 (26) | 13 (21) | 28 (36) | 24 (36)
Peripheral sensory neuropathy (Nervous system disorders) | 17 (17) | 20 (20) | 21 (29) | 18 (23) | 38 (46) | 38 (43)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 5 (5) | 3 (4) | 5 (5) | 4 (5)
Anxiety (Psychiatric disorders) | 7 (9) | 8 (8) | 8 (8) | 2 (2) | 15 (17) | 10 (10)
Insomnia (Psychiatric disorders) | 45 (48) | 45 (49) | 18 (20) | 12 (12) | 63 (68) | 57 (61)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 23 (23) | 12 (14) | 10 (13) | 33 (36) | 33 (36)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 5 (5) | 3 (3) | 7 (7) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 7 (7) | 14 (14) | 11 (11) | 31 (32) | 18 (18)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 8 (8) | 7 (8) | 9 (10) | 20 (21) | 17 (18)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 28 (55) | 29 (58) | 10 (11) | 3 (3) | 38 (66) | 32 (61)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 9 (9) | 4 (4) | 14 (14) | 10 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 3 (3) | 10 (11) | 5 (5) | 22 (24) | 8 (8)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 5 (5) | 2 (2) | 7 (7) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (9) | 5 (5) | 3 (4) | 11 (11) | 10 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (24) | 16 (17) | 30 (33) | 28 (32) | 52 (57) | 44 (49)
Dry skin (Skin and subcutaneous tissue disorders) | 20 (21) | 11 (11) | 13 (14) | 4 (5) | 33 (35) | 15 (16)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4) | 6 (13) | 6 (7) | 12 (19) | 10 (11)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 67 (74) | 57 (68) | 5 (5) | 10 (10) | 72 (79) | 67 (78)
Pruritus (Skin and subcutaneous tissue disorders) | 59 (69) | 23 (28) | 16 (22) | 6 (7) | 75 (91) | 29 (35)
Rash (Skin and subcutaneous tissue disorders) | 45 (51) | 30 (36) | 22 (27) | 12 (13) | 67 (78) | 42 (49)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (8) | 5 (6) | 6 (8) | 2 (2) | 13 (16) | 7 (8)
Deep vein thrombosis (Vascular disorders) | 6 (6) | 8 (8) | 5 (5) | 4 (4) | 11 (11) | 12 (12)
Hypertension (Vascular disorders) | 25 (29) | 30 (38) | 8 (9) | 9 (15) | 33 (38) | 39 (53)
Hypotension (Vascular disorders) | 21 (21) | 9 (10) | 8 (9) | 9 (9) | 29 (30) | 18 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03221426/Prot_SAP_000.pdf